CLINICAL TRIAL: NCT05404958
Title: Systems Analysis and Improvement Approach to Improve Integration of HIV Prevention and Treatment Services
Acronym: FP HIV SCALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, McKenna Eastment, Assistant Professor: Department of Medicine, Division of Allergy & Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014745; GRANT13455302 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-02

CONDITIONS: Hiv
Keywords: HIV prevention and treatment; Family planning; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial enrolling family planning clinics. "Participants" are FP clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention clinics that implement the Systems Analysis and Improvement Approach (Experimental): Mombasa County public health staff will facilitate SAIA
  Interventions: Other: Systems Analysis and Improvement Approach (SAIA)
- Usual procedures (No Intervention)

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach (SAIA) — What is SAIA? It is a 5-step cycle that is repeated every 4-6 weeks for continuous quality improvement, implemented by Kenyan public health workforce and FP clinic staff, and monitored by Mombasa DOH.
  Step 1: Understanding the cascade from FP clinic enrollment to HIV testing to linkage to treatment and prevention services.
  Step 2: Use process mapping to identify modifiable bottlenecks. Step 3: Define and implement workflow adaptations to eliminate modifiable bottlenecks.
  Step 4: Monitor change in performance. Step 5: Repeat the analysis and improvement cycle (steps 1-4).
  Arms: Intervention clinics that implement the Systems Analysis and Improvement Approach

SUMMARY:
East and Southern Africa is home to 6.2% of the world's population but includes 54% of all people living with HIV (PLWH). In this region, three out of five PLWH are women, and there is a particularly high burden of HIV amongst adolescent girls and young women (AGYW). Over half of African women use family planning (FP) services. Integration of HIV prevention and treatment with FP services holds promise for supporting progress toward the UNAIDS 95-95-95 targets for testing, treatment, and prevention. Nonetheless, integration of even basic HIV prevention and treatment services into FP clinics remains low and how best to integrate these services is still unknown. In a previous trial, the Systems Analysis and Improvement Approach (SAIA), was an effective implementation strategy for improving HIV counseling and testing in a small selection of FP clinics in Mombasa County, Kenya when delivered by research staff. SAIA incorporates a cascade analysis tool, sequential process flow mapping, and cycles of micro-intervention development, implementation, and assessment to improve a care cascade. More data is needed to understand if SAIA is effective for also improving linkage to HIV care and screening and linkage to pre-exposure prophylaxis (PrEP) in FP clinics when SAIA is delivered at scale by Kenyan public health workforce. The first objective of this study is to conduct a cluster-randomized trial evaluating the effectiveness of SAIA versus control (usual procedures with no specific intervention) for increasing HIV counseling, testing, linkage to HIV care, and screening and linkage to PrEP in new FP clients and new and returning AGYW clients. There will be a particular focus on the HIV prevention and treatment of AGYW in this study and any AGYW presenting for FP care will be prioritized. Quantitative and qualitative data will be analyzed using the RE-AIM framework to evaluate the program's Reach, Effectiveness, Adoption, Implementation, and Maintenance. To understand how SAIA could be integrated into national Ministry of Health policies and programs, activity-based costing will be conducted to estimate the budget and program impacts of SAIA, scaled to a County level, from a Ministry of Health perspective. It is hypothesized that compared to control, SAIA will be effective at increasing HIV counseling, HIV testing, linkage to HIV care, and screening and linkage to PrEP for new FP clients and all new and returning AGYW FP clients when delivered at scale by Kenyan public health staff. The implementation evaluation, costing, and budget impact analysis will establish a road map for national-level implementation, positioning Kenya as a global leader in integrating FP/HIV services.

DETAILED DESCRIPTION:
AIM 1: To conduct a cluster-randomized trial evaluating the effectiveness of SAIA versus control (usual procedures) for increasing HIV counseling, testing, linkage to care, and screening and linkage to PrEP in new FP clients and new and returning AGYW clients. Quantitative and qualitative data will be analyzed using the RE-AIM framework (21).

1a) Reach: Proportion of intervention arm health facility clients' reached with the intervention

1b) Effectiveness: Compare the effectiveness of SAIA vs. control for increasing rates of HIV counseling, testing, linkage to care, and screening and linkage to PrEP in new FP clients and new and returning AGYW clients

1c) Adoption: Proportion of clinics adopting SAIA; adoption determinants identified using the Implementation Research Logic Model (IRLM) (22) and Organizational Readiness for Implementing Change (ORIC) scale (23)

1d) Implementation: Proportion of FP clinics implementing SAIA with high fidelity at 12 months and at 24 months; barriers and facilitators of implementation at scale by County DOH personnel will be explored using constructs from the Consolidated Framework for Implementation Research (CFIR) and the IRLM (24)

1e) Maintenance: Proportion of FP clinics maintaining SAIA at 12 months and 24 months after introduction AIM 2: To estimate the incremental cost and budget and program impacts of SAIA from a County DOH perspective. We will conduct activity-based costing and develop budget impact scenarios based on SAIA's adoption.

ELIGIBILITY:
Inclusion Criteria:

FP clinics:

-All FP clinics that receive County-supplied FP products will be eligible to participate.

FP clinic managers and staff:

-Any FP clinic manager that is 18 years and older is eligible to be interviewed. -These clinic managers can be male or female.

Kenyan public health staff:

* Any Kenyan public health staff that is 18 years and older is eligible to be interviewed.
* These public health staff can be male or female.

Exclusion Criteria:

FP clinics:

* Any clinics that are expected to close within the next year at the time of study initiation
* 12 facilities that participated as SAIA intervention facilities in our small-scale trial where the intervention was led by research staff.

FP clinic managers and staff: No exclusion criteria Kenyan public health staff: No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness HIV counseling | Months 1-24
  Proportion of new FP clients and all AGYW clients that are counseled for HIV out of the total new FP clients and AGYW in intervention vs control clinics
Effectiveness HIV testing | Months 1-24
  Proportion of new FP clients and all AGYW tested for HIV out of the total new FP clients and all AGYW who are eligible to be tested in intervention vs control clinics
Effectiveness Linked to HIV care | Months 1-24
  Proportion of HIV-seropositive new FP clients and all HIV-seropositive AGYW clients linked to comprehensive HIV care out of all HIV-seropositive new FP clients and all HIV-seropositive AGYW clients in intervention vs control clinics
Effectiveness Screening for PrEP | Months 1-24
  1. Proportion of new FP clients and all AGYW clients screened for PrEP out of all new FP clients and all AGYW clients who were counseled for HIV in intervention vs control clinics
Effectiveness linkage to PrEP | 1-24 months
  Proportion of new FP clients and all AGYW clients who are eligible for PrEP who are linked to PrEP out of all new FP clients and all AGYW who are eligible for PrEP in intervention vs control clinics

CONTACTS AND LOCATIONS:
Overall Officials: McKenna Eastment, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- FP Clinics in Mombasa County, Mombasa, Kenya